CLINICAL TRIAL: NCT07122947
Title: Surveillance Trial of the Apple Watch in Reliable Burden Assessment in Unseen Recurrence of Surgically Treated Atrial Fibrillation (STARBURST-AF)
Brief Title: Surveillance Trial of the Apple Watch in Reliable Burden Assessment in Unseen Recurrence of Surgically Treated AF
Acronym: STARBURST-AF
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Marc Gillinov, MD, Principal Investigator, The Cleveland Clinic
Other Study IDs: 25-458
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
Keywords: Wearable; Apple Watch; Atrial Fibrillation; Arrhythmia; Zio Patch; Ambulatory Rhythm Monitoring
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Photoplethysmography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Apple Watch: AFib History — The Apple Watch AFib History feature uses PPG pulse rhythm data to detect and quantify the burden of atrial fibrillation.
  Other Names: Apple Watch Series 10; Photoplethysmography (PPG) Pulse Rhythm Monitoring
Device: Zio Patch — The 14-day Zio Patch monitoring device (iRhythm Technologies, Inc., San Francisco, CA) uses continuous ambulatory ECG monitoring to quantify the burden of atrial fibrillation.
  Other Names: iRhythm Zio Patch; Continuous Ambulatory ECG Monitoring

SUMMARY:
This is a prospective multicenter clinical study comparing the efficacy of the Apple Watch AFib History tool to the iRhythm Zio Patch monitoring device in quantifying atrial fibrillation (AF) burden after surgical ablation. Patients with AF and mitral valve (MV) disease who undergo a Cox-Maze IV procedure concomitant to MV surgery will be evaluated at serial timepoints for up to 1 year postoperatively. The trial will be conducted in the United States at the Cleveland Clinic in Cleveland, OH and at the Washington University School of Medicine in St. Louis, MO.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the accuracy of current wearable technology using the Apple Watch AFib History tool, relative to ambulatory electrocardiogram (ECG) monitoring using the Zio Patch, for quantifying AF burden after surgical ablation. AF burden will be measured as a weekly estimate, defined as the percentage of time in AF over the prior seven consecutive days. This assessment will occur at 3 months, 6 months, and 1 year postoperatively.

This is a paired study design in which each subject will receive both the investigational device (Apple Watch) and reference device (Zio Patch) concurrently. The study population includes adults over the age of 22 years with a documented history of AF and MV disease undergoing elective MV surgery with concomitant Cox-Maze IV surgical ablation. All participants must be able to provide informed consent and adhere to the study follow-up schedule. Participants who meet the eligibility criteria will be enrolled on a rolling basis. Pre-surgical questionnaires, including Patient-Reported Outcomes Measurement Information System (PROMIS-10), MacNew, and Atrial Fibrillation Severity Scale (AFSS) surveys will be implemented at baseline and serial follow-up.

The monitoring period will be conducted in phases during serial follow-up at 1 month, 3 months, 6 months, and 1 year postoperatively. The Apple Watch will be worn postoperatively for the study duration. Participants will be instructed to charge the device overnight. The Zio Patch 14-day ambulatory ECG monitor will be applied at the following study timepoints: 3 months, 6 months, and 1 year postoperatively. Participants will be instructed to wear the Apple Watch concurrently during Zio Patch monitoring periods, as well as in the interval between visits.

At each follow-up visit (1 month, 3 months, 6 months, and 1 year), participants will undergo standardized evaluations, including a physical exam and the administration of the same standardized questionnaires. Comparative data from the Apple Watch and Zio Patch will be analyzed at the 3 months, 6 months, and 1 year visits.

ELIGIBILITY:
Inclusion Criteria:

* 22 years of age or older
* Documented or current history of atrial fibrillation (paroxysmal, persistent, or long-standing persistent)
* Undergoing elective mitral valve surgery (repair or replacement) with concomitant surgical ablation using a Cox-Maze IV lesion set and left atrial appendage occlusion procedure, with and without concomitant tricuspid valve procedure (repair or replacement)
* Use or access to Apple iPhone
* Willing and able to provide informed consent and wear both the Apple Watch and Zio Patch at pre-specified intervals for the duration of the study period
* Willing and able to participate in long-term follow up including study visits and surveys

Exclusion Criteria:

* Presence of a cardiac pacemaker
* Heart failure with reduced ejection fraction (<40%)
* Concomitant aortic valve replacement or coronary artery bypass graft
* Personal or family history of adhesive skin allergies to adhesives or hydrogels
* Tattoos located on the skin of the wrist or forearm where the Apple Watch will be placed
* Pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>22 years) with a documented history of atrial fibrillation and mitral valve disease who undergo surgical ablation with a Cox-Maze IV concomitant to elective mitral valve surgery.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AF burden | From enrollment to 1 year postoperatively
  This will be measured by comparing the weekly AF burden estimates from the Apple Watch AF History feature to the Zio Patch ambulatory ECG monitoring device. Weekly AF burden is defined as the percentage of time in AF over the prior seven consecutive days and will be measured at 3 months, 6 months, and 1 year postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gillinov, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No